CLINICAL TRIAL: NCT05576103
Title: Longitudinal Prospective Study of Neurocognitive Outcomes and Multimodal Quantitative Neuroimaging Outcomes in Primary Brain Tumor Patients Receiving Brain Radiotherapy
Brief Title: Longitudinal Prospective Study of Neurocognition & Neuroimaging in Primary BT Patients
Status: Recruiting | Type: Observational
Sponsor: Jona Hattangadi-Gluth (Other)
Responsible Party: Sponsor-Investigator, Jona Hattangadi-Gluth, Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Other Study IDs: 131457
Record Dates: First submitted 2022-10-07; First posted 2022-10-12 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Primary Brain Tumor; Glioma; Meningioma; Schwannoma
MeSH Terms: conditions — Brain Neoplasms; Glioma; Meningioma; Neurilemmoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary brain tumour patients receiving RT: Primary brain tumor patients are screened at time of consultation for this observational study, and the study population is diverse across sex/gender, and racial/ethnic groups.

SUMMARY:
In this proposal, the investigators introduce a novel, translational study to prospectively examine primary brain tumor patients undergoing fractionated radiation therapy to the brain. Quantitative neuroimaging, radiation dose information, and directed neurocognitive testing will be acquired through this study to improve understanding of cognitive changes associated with radiation dosage to non-targeted tissue, and will provide the basis for evidence-based cognitive- sparing brain radiotherapy.

DETAILED DESCRIPTION:
Background: Fractionated radiation therapy (RT) is a mainstay in the treatment of primary and metastatic brain tumors. However, RT to the brain is associated with an inevitable decline in neurocognitive function in up to 90% of patients who survive more than 6 months after irradiation. Radiation to the brain results in an inevitable decline in neurocognitive function, mediated by tissue injury to white matter, cortex and subcortical areas. With quantitative magnetic resonance imaging (MRI) techniques, investigators can directly and non-invasively measure such changes.

Objective/Hypothesis:

The purpose of this study is to examine radiation-induced imaging changes in normal brain tissue over time in primary brain tumor patients, and correlate these with neurocognitive outcomes. The overarching goal is to better identify sensitive brain regions so that future radiation techniques can be optimally designed to mitigate collateral damage.

Specific Aims:

1. To identify microstructural changes in subcortical white matter, hippocampus, and cortex associated with quantified regional exposure to fractionated brain radiotherapy using advanced quantitative neuroimaging imaging
2. To identify changes in neurocognitive functioning in primary brain tumor patients after brain radiotherapy

Study Design:

The investigators will prospectively enroll primary brain tumor patients undergoing fractionated partial brain radiation therapy. Patients will undergo volumetric and diffusion brain MRI (per clinical standard-of-care) and a neurocognitive battery of tests at baseline (pre-treatment), 3 months, 6 months, and 12 months post-treatment. Clinical data including age, gender, educational status, tumor size and histology, steroid use, antiepileptic drug use and chemotherapy will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years or older
2. Karnofsky performance status (KPS) ≥70
3. Life expectancy of ≥1 year
4. Primary brain tumor patients who will receive fractionated partial brain RT
5. Able to complete neurocognitive assessments

Exclusion Criteria:

1. Inability to undergo MRI with contrast
2. Prior brain RT

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary brain tumor patients
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Longitudinal changes in imaging biomarker volume (cc) from volumetric MR imaging | baseline (pre-treatment), 3 months, 6 months, 12 months post-treatment
  To measure longitudinal changes in volume (cc) from volumetric MR imaging
Longitudinal changes in imaging biomarker mean diffusivity (MD) in white matter from DTI imaging | baseline (pre-treatment), 3 months, 6 months, 12 months post-treatment
  To measure longitudinal changes in MD (mm squared/second) from DTI imaging
Longitudinal changes in imaging biomarker fractional anisotropy (FA) in white matter from DTI imaging | baseline (pre-treatment), 3 months, 6 months, 12 months post-treatment
  To measure longitudinal changes in FA (unitless index between 0 and 1) from DTI imaging
Change in Memory after RT | baseline (pre-treatment), 3 months, 6 months, 12 months post-treatment
  To evaluate the change from baseline to post-RT verbal memory performance when performing fractionated partial brain RT. Verbal memory outcomes and measurements include: Hopkins Verbal Learning Test-Revised (HVLT-R)-Immediate, Delayed Recall. Brief Visuospatial Memory Test-Revised (BVMT-R)- Total, Delayed Recall
  Scale of scores is:
  Hopkins Verbal Learning Test-Revised (HVLT-R)-Immediate, Delayed Recall: 0-36 for Immediate, 0-12 for Delayed. For both tests, higher scores indicate better performance.
  Brief Visuospatial Memory Test-Revised (BVMT-R)- Total, Delayed Recall: l: 0-36 for Immediate, 0-12 for Delayed.
  For both tests, higher scores indicate better performance.
Change in Executive Functioning after RT | baseline (pre-treatment), 3 months, 6 months, 12 months post-treatment
  To evaluate the change from baseline to post-RT executive functioning performance when performing fractionated partial brain RT. Executive functioning outcomes and measurements include: Controlled Oral Word Association Test (COWA): letter fluency, Trail Making Test Part B (TMT-B).
  Scale of scores is:
  Controlled Oral Word Association Test (COWA): letter fluency: 0- no upper limit. Higher score indicates better performance Trail Making Test Part B (TMT-B): 0-240. Higher score indicates poorer performance
Change in Attention/Processing Speed after RT | baseline (pre-treatment), 3 months, 6 months, 12 months post-treatment
  To evaluate the change from baseline to post-RT Attention/Processing Speed performance when performing fractionated partial brain RT. Attention/Processing Speed outcomes and measurements include: Trail Making Test Part A (TMT-A)
  Scale of scores is:
  Trail Making Test Part A (TMT-A): 0-240. Higher score indicates poorer performance.
Change in Language functioning after RT | baseline (pre-treatment), 3 months, 6 months, 12 months post-treatment
  To evaluate the change from baseline to post-RT Language performance when performing fractionated partial brain RT in patients with primary brain tumor. Language outcomes and measurements include: Boston Naming Test (BNT), Controlled Oral Word Association Test (COWA): category fluency
  Scale of scores is:
  Boston Naming Test (BNT): 0-60 Controlled Oral Word Association Test (COWA): category fluency: 0-no upper limit.
  For both tests, higher score indicates better performance.
Change in Fine Motor Skills after RT | baseline (pre-treatment), 3 months, 6 months, 12 months post-treatment
  To evaluate the change from baseline to post-RT Fine Motor Skills performance when performing fractionated partial brain RT in patients with primary brain tumor. Fine Motor Skills outcomes and measurements include:
  Trail Making Test Motor Speed; Grooved Pegboard Test
Change in health-related quality of life (hrQoL) from baseline to 5 years after RT | baseline (pre-treatment), 3 months, 6 months, 12 months post-treatment
  To evaluate the change from baseline to post-RT health-related quality of life (hrQoL) when performing fractionated partial brain RT in patients with primary brain tumor. Quality of life outcomes and measurements include: Beck Depression inventory II (BDI II), Beck Anxiety Inventory (BAI) and FACT-BR (Functional Assessment of Cancer Therapy - Brain).
  FACT-BR (Functional Assessment of Cancer Therapy - Brain) higher scores on each subscale indicate greater hrQoL.

CONTACTS AND LOCATIONS:
Locations (1):
- Moores Cancer Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Greene-Schloesser D, Robbins ME. Radiation-induced cognitive impairment--from bench to bedside. Neuro Oncol. 2012 Sep;14 Suppl 4(Suppl 4):iv37-44. doi: 10.1093/neuonc/nos196. PMID 23095829
- [Background] Huynh-Le MP, Tibbs MD, Karunamuni R, Salans M, Tringale KR, Yip A, Connor M, Simon AB, Vitzthum LK, Reyes A, Macari AC, Moiseenko V, McDonald CR, Hattangadi-Gluth JA. Microstructural Injury to Corpus Callosum and Intrahemispheric White Matter Tracts Correlate With Attention and Processing Speed Decline After Brain Radiation. Int J Radiat Oncol Biol Phys. 2021 Jun 1;110(2):337-347. doi: 10.1016/j.ijrobp.2020.12.046. Epub 2021 Jan 4. PMID 33412257
- [Background] Salans M, Tibbs MD, Karunamuni R, Yip A, Huynh-Le MP, Macari AC, Reyes A, Tringale K, McDonald CR, Hattangadi-Gluth JA. Longitudinal change in fine motor skills after brain radiotherapy and in vivo imaging biomarkers associated with decline. Neuro Oncol. 2021 Aug 2;23(8):1393-1403. doi: 10.1093/neuonc/noab017. PMID 33543265
- [Background] Tibbs MD, Huynh-Le MP, Karunamuni R, Reyes A, Macari AC, Tringale KR, Salans M, Yip A, Liu E, Simon A, McDonald CR, Hattangadi-Gluth JA. Microstructural Injury to Left-Sided Perisylvian White Matter Predicts Language Decline After Brain Radiation Therapy. Int J Radiat Oncol Biol Phys. 2020 Dec 1;108(5):1218-1228. doi: 10.1016/j.ijrobp.2020.07.032. Epub 2020 Jul 23. PMID 32712255
- [Background] Tringale KR, Nguyen TT, Karunamuni R, Seibert T, Huynh-Le MP, Connor M, Moiseenko V, Gorman MK, Marshall A, Tibbs MD, Farid N, Simpson D, Sanghvi P, McDonald CR, Hattangadi-Gluth JA. Quantitative Imaging Biomarkers of Damage to Critical Memory Regions Are Associated With Post-Radiation Therapy Memory Performance in Brain Tumor Patients. Int J Radiat Oncol Biol Phys. 2019 Nov 15;105(4):773-783. doi: 10.1016/j.ijrobp.2019.08.003. Epub 2019 Aug 10. PMID 31408667
- [Background] Seibert TM, Karunamuni R, Bartsch H, Kaifi S, Krishnan AP, Dalia Y, Burkeen J, Murzin V, Moiseenko V, Kuperman J, White NS, Brewer JB, Farid N, McDonald CR, Hattangadi-Gluth JA. Radiation Dose-Dependent Hippocampal Atrophy Detected With Longitudinal Volumetric Magnetic Resonance Imaging. Int J Radiat Oncol Biol Phys. 2017 Feb 1;97(2):263-269. doi: 10.1016/j.ijrobp.2016.10.035. Epub 2016 Oct 31. PMID 28068234
- [Background] Meyers CA, Rock EP, Fine HA. Refining endpoints in brain tumor clinical trials. J Neurooncol. 2012 Jun;108(2):227-30. doi: 10.1007/s11060-012-0813-8. Epub 2012 Mar 27. PMID 22451194
- [Derived] Connor M, Salans M, Karunamuni R, Unnikrishnan S, Huynh-Le MP, Tibbs M, Qian A, Reyes A, Stasenko A, McDonald C, Moiseenko V, El-Naqa I, Hattangadi-Gluth JA. Fine Motor Skill Decline After Brain Radiation Therapy-A Multivariate Normal Tissue Complication Probability Study of a Prospective Trial. Int J Radiat Oncol Biol Phys. 2023 Nov 1;117(3):581-593. doi: 10.1016/j.ijrobp.2023.04.033. Epub 2023 May 6. PMID 37150258